CLINICAL TRIAL: NCT05038631
Title: Managed Access Programs for LEE011, Ribociclib
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011A2408
Record Dates: First submitted 2021-08-18; First posted 2021-09-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: MAP; Manage access program; Breast Cancer; CLEE011; Ribociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Ribociclib — Patients receive ribociclib
  Other Names: LEE011

SUMMARY:
The purpose of this registration is to list Managed Access Programs (MAPs) related to LEE011, Ribociclib

DETAILED DESCRIPTION:
CLEE011A2408 - No longer available - Managed Access Program (MAP) Cohort to provide access to ribociclib (LEE011, Kisqali®), for locally advanced or metastatic cancer resistant or refractory to available treatment options and candidate for therapy with a CDK inhibitor (including tumors with D-cyclin-CDK4/6-INK4a-Rb pathway abnormalities)

CLEE011A2006M - Available - Managed Access Program (MAP) Cohort to provide access to Ribociclib for patients diagnosed with early-stage HR+HER2 (stages II and III) - breast cancer requiring adjuvant treatment with an ET based regimen

ELIGIBILITY:
Inclusion Criteria:

1. An independent request was received from a licensed physician.
2. The patient has a serious or life-threatening disease or condition and there is no comparable or satisfactory alternative therapy available for diagnosis, monitoring, or treatment.
3. The patient is not eligible or able to enroll in a clinical trial or continue participation in such trial.
4. There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
5. The patient must meet any other medical criteria established by the medical experts responsible for the product or by the health authority in the country of request (as applicable).
6. Provision of the product will not interfere with the initiation, conduct, or completion of a Novartis clinical trial or overall development program.
7. Managed Access provision is allowed per local laws/regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult